CLINICAL TRIAL: NCT01741285
Title: Effects Of Extra-fine Particle HFA-becLomethasone (HFA-QVAR) Versus Course Particle Treatment In Smokers and Ex-smokers With Asthma
Brief Title: Effects of QVAR in Smokers With Asthma
Acronym: OLiVIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Teva Pharma (Industry)
Responsible Party: Principal Investigator, Maarten van den Berge, Chest Physician, University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20122011
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: Asthma; Adenosine; Small airways; Smokers; Ex-smokers
MeSH Terms: conditions — Asthma; Smoking Cessation | interventions — Beclomethasone; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fluticasone (Active Comparator): Two weeks treatment with HFA-Fluticasone 250 microgram twice daily
  Interventions: Drug: Beclomethasone (QVAR); Drug: Beclomethasone (Clenil)
- Clenil (Active Comparator): Two weeks treatment with HFA-Clenil 200 microgram 2 inhalations twice daily.
  Interventions: Drug: Beclomethasone (QVAR); Drug: Fluticasone
- QVAR (Experimental): Two weeks treatment with QVAR 2 times 100 microgram twice daily
  Interventions: Drug: Beclomethasone (Clenil); Drug: Fluticasone

INTERVENTIONS:
Drug: Beclomethasone (QVAR) — Small particle treatment
  Other Names: QVAR
  Arms: Clenil; Fluticasone
Drug: Beclomethasone (Clenil) — Course particle beclomethasone
  Other Names: Clenil
  Arms: Fluticasone; QVAR
Drug: Fluticasone — Course particle treatment
  Other Names: Flixotide
  Arms: Clenil; QVAR

SUMMARY:
We hypothesize that extra-fine particle treatment with HFA-QVAR will be superior in improving small airways dysfunction, especially in ex-smokers and smokers with asthma.

To investigate this, we will perform a study comparing the efficacy of extra-fine particle HFA-QVAR 200 µg b.i.d. to an equipotent dose of course particle HFA-beclomethasone (HFA-Clenil) 400 µg b.i.d. and with coarse particle HFA-fluticasone (GSK) 250 µg in ex-smokers and smokers with asthma.

Study design: This study will be an open-label, randomised, three-way cross-over, two-center study. 20 smokers and 20 ex-smokers with asthma will receive the following treatments for two weeks:

DETAILED DESCRIPTION:
Rationale:

Thus far, most clinical studies investigating the effects of inhaled corticosteroids (ICS) in asthma have concentrated on non-smoking asthmatics. However, a considerable proportion of asthma patients smokes. Cigarette smoke consists of ultra-fine particles with a diameter between 0.1 and 1 µm and therefore reaches even the smallest airways. In line with this, it has been reported that smoking is associated with small airways dysfunction. The latter may help to explain the observation that treatment with course particle inhaled corticosteroids is less effective in smokers with asthma. Recently, extra-fine particle aerosols such as hydrofluoroalkane-beclomethasone (HFA-QVAR) have become available for the treatment of asthma, which are more likely to reach the smaller airways. Based on the above, we hypothesize that extra-fine particle treatment with HFA-QVAR will be superior in improving small airways dysfunction, especially in ex-smokers and smokers with asthma.

Objective: To perform a study comparing the efficacy of extra-fine particle HFA-QVAR 200 µg b.i.d. to an equipotent dose of course particle HFA-beclomethasone (HFA-Clenil) 400 µg b.i.d. and with coarse particle HFA-fluticasone (GSK) 250 µg in ex-smokers and smokers with asthma.

Study design:

This study will be an open-label, randomised, three-way cross-over, two-center study. 20 smokers and 20 ex-smokers with asthma will receive the following treatments for two weeks:

Treatment period A: 2-week treatment with HFA-QVAR (TEVA Pharma) 200 μg b.i.d. Treatment period B: 2-week treatment with HFA-Clenil (Chiesi) 400 μg b.i.d. Treatment period C: 2-week treatment with HFA-Fluticasone (GlaxoSmithKline) 250 μg b.i.d.

Study population:

20 smokers and 20 ex-smokers with asthma, aged 18-65 years, will receive the following treatments for two weeks:

Intervention (if applicable):

A: 2-week treatment with HFA-QVAR (TEVA) 200 μg b.i.d. B: 2-week treatment with HFA-Clenil (Chiesi) 400 μg b.i.d. C: 2-week treatment with HFA-Fluticasone (GlaxoSmithKline) 250 μg b.i.d.

Main study parameters/endpoints: The primary end-parameter is the decrease in peripheral airways resistance (R5-R20) at the provocative dose of small particle adenosine causing the Forced Expiratory Volume in one second (FEV1) to drop with 20%. The co-primary end-parameter is the PD20 small particle adenosine.

All patients will attend 7 visits to the outpatient clinic. At baseline and after treatment, the following investigations will be performed: PC20AMP, PD20 small particle adenosine, spirometry, IOS, body plethysmography, blood collection, filling in of questionnaires, and nasal epithelial brushings.

ELIGIBILITY:
3.1 Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Males and females with a doctor's diagnosis of asthma
* Age between 18 and 65 years
* Current- and ex-smokers with ≥ 5 packyears.
* Drop in FEV1 > 20% after provocation with small particle adenosine < 20 mg at visit 1.

3.2 Exclusion criteria

A subject who meets any of the following criteria will be excluded from participation in this study:

* An asthma exacerbation during the last 6 weeks or upper respiration tract infection during the last 4 weeks prior to inclusion in the study.
* Severe airway obstruction at baseline, FEV1 < 50% of predicted or < 1.2 liter.
* Physician diagnosed predominant COPD or any other pulmonary disease that could influence the study results as judged by the investigator.
* Pregnant or lactating women.
* Females of childbearing potential without an efficient contraception unless they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or the use of one or more of the following acceptable methods of contraception:

  1. Surgical sterilization (e.g. bilateral tubal ligation, hysterectomy).
  2. Hormonal contraception (implantable, patch, oral, injectable).
  3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/cream/suppository.
  4. Continuous abstinence. Periodic abstinence (e.g. calendar, ovulation, symptom-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Reliable contraception should be maintained throughout the study and for 30 days after study drug discontinuation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
PD20 Adenosine | This measurement will be performed at baseline and after two weeks treatment with either QVAR, Clenil or Fluticasone
  The primary end-parameter is the PD20 small particle adenosine. The co-primary objective (only in case of non-inferiority of QVAR on the primary objective) will be: Reduction in peripheral airways resistance (R5-R20) measured with IOS at the provocative dose of small particle adenosine causing the FEV1 to drop with 20% (PD20).

SECONDARY OUTCOMES:
Symptoms and Peakflow | This measurement will be performed at baseline and after two weeks treatment with either QVAR, Clenil or Fluticasone
  Twice daily symptoms (including night-time symptoms) and peakflow (PEF).
Airway resistance | This measurement will be performed at baseline and after two weeks treatment with either QVAR, Clenil or Fluticasone
  Resistance (R5, R20, R5-R20) and Reactance at 5 Herz (X5) with IOS.
Spirometry | This measurement will be performed at baseline and after two weeks treatment with either QVAR, Clenil or Fluticasone
  FEF25, FEF50, FEF75, FEF25-75, PEF, FEV1, FEV1/FVC, FVC/SVC
Body Plethysmography | This measurement will be performed at baseline and after two weeks treatment with either QVAR, Clenil or Fluticasone
  RV (%predicted), TLC, RV/TLC (%), FRC, FRC/TLC (%), FRC/TLC (%predicted), IC, RV/TLC %predicted
Peripheral blood | This measurement will be performed at baseline and after two weeks treatment with either QVAR, Clenil or Fluticasone
  cell differential counts, DNA, PBMC's, serum.
Delta FVC during PD20 small particle adenosine. | This measurement will be performed at baseline and after two weeks treatment with either QVAR, Clenil or Fluticasone
Questionnaires | This measurement will be performed at baseline and after two weeks treatment with either QVAR, Clenil or Fluticasone
  ACQ, BHQ, CCq
Multiple Breath Washout Analysis | This measurement will be performed at baseline and after two weeks treatment with either QVAR, Clenil or Fluticasone
  If possiboe this measurement will be performed.
Nasal brushing | This measurement will be performed at baseline and after two weeks treatment with either QVAR, Clenil or Fluticasone
  Genome-wide gene (mRNA and microRNA) expression and DNA methylation in nasal brushings

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van den Berge, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Cox CA, Boudewijn IM, Vroegop SJ, Schokker S, Lexmond AJ, Frijlink HW, Hagedoorn P, Vonk JM, Farenhorst MP, Ten Hacken NHT, Kerstjens HAM, van den Berge M. Associations of AMP and adenosine induced dyspnea sensation to large and small airways dysfunction in asthma. BMC Pulm Med. 2019 Jan 28;19(1):23. doi: 10.1186/s12890-019-0783-0. PMID 30691429